CLINICAL TRIAL: NCT02454673
Title: Approximation to the Therapeutic Individualization in Patients With Locally Advanced Gastric and Gastroesophageal Cancer Through Modelling and Generation of Predictive Gene Signatures
Brief Title: Therapeutic Individualization for Patients With Locally Advanced Gastric and Gastroesophageal Cancer
Status: Completed | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: CUN-GCNMEM
Record Dates: First submitted 2015-05-22; First posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-03

CONDITIONS: Gastric Cancer; Effects of Chemotherapy; Surgery
Keywords: Radiotherapy; Neoadjuvant therapy; Pharmacodynamics; Pharmacokinetics; Nonlinear Dynamics
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Surgical specimen with potential for extraction of DNA.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: * 3-4 cycles of preoperative chemotherapy
  * Surgery
- Group B: * 3-4 cycles of induction chemotherapy
  * Radiotherapy with concurrent chemotherapy for 5 weeks
  * Surgery

SUMMARY:
The purpose of this study is to evaluate whether the R0 rate, pathological response degree, patterns of recurrence and long-term outcomes may be initially predicted in patients with locally advanced gastroesophageal junction and gastric cancer treated with a neoadjuvant approach and salvage surgery.

DETAILED DESCRIPTION:
Patients with locally advanced gastroesophageal junction and gastric cancer with T3-4 and/or N+ are included. Initially, patients are diagnosed by computerized tomography scan and endoscopic ultrasound. The neoadjuvant strategy consisted of 3-4 cycles of preoperative chemotherapy (group A) or 3-4 courses of induction chemotherapy followed by concurrent chemoradiotherapy (group B). Chemoradiotherapy comprised weekly chemotherapy concurrently with daily external beam radiotherapy up to 45 Gy). Surgery is scheduled 4 to 6 weeks after the end of CRT. Pathological response is graded according to the Becker criteria. Statistical analysis is performed IBM SPSS v20. Nonlinear mixed effects (NLME) modelling is applied to evaluate the impact of dynamic changes in tumor size, neutrophil lymphocyte ratio (NLR) and platelet lymphocyte ratio (PLR) on the clinical outcome of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the stomach or gastroesophageal cancer
* Age ≥18 years old
* Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-1
* Body mass index ≥ 18
* No prior chemotherapy or chemoradiotherapy
* TNM stage of T3-T4 and/or positive regional lymph nodes (N+) by endoscopic ultrasound or computed tomography (CT)
* No evidence of metastasis (M0)
* Adequate hematological, liver and renal functions (ALT and AST≤2.5 UNL, total bilirubin ≤1.5 UNL, and serum creatinine ≤1.5 UNL)

Exclusion Criteria:

* Patients with previous (less than 10 years) or current history of malignant neoplasms, except for curatively treated
* Patients with evidence of severe or uncontrolled systemic disease
* Medically unfit for chemotherapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced adenocarcinoma gastric cancer for a neoadjuvant protocol consisting of preoperative chemotherapy or induction chemotherapy, chemoradiotherapy and salvage surgery. Patients must have a medically fit condition to complete the protocol.
  Initial staging comprises a thoracic and abdominal computerised tomography scan, endoscopic ultrasound endoscopy (EUS), biopsy and blood test including blood cell count, hepatic and renal function.
  Radiological and endoscopic evaluations are performed at baseline and at the completion of chemotherapy and chemoradiotherapy.
  Blood tests are acquired at baseline, before each chemotherapy course and concurrently with evaluations. Blood tests are also obtained during follow-up and at the time progression.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Overall Survival | From date of diagnosis until death, assessed up to 10 years
  Overall survival was defined as the period from diagnosis until death (from any cause). Nonlinear mixed effects population modelling to evaluate the impact in clinical outcome of dynamic markers as tumor size, neutrophil lymphocyte ratio (NLR) and platelet lymphocyte ratio (PLR).
Disease Free Survival | From date of diagnosis until treatment failure, assessed up to 10 years
  DFS was defined as the time from diagnosis to the first date of local or distant cancer. Nonlinear mixed effects population modelling to evaluate the impact in clinical outcome of dynamic markers as tumor size, neutrophil lymphocyte ratio (NLR) and platelet lymphocyte ratio (PLR).

SECONDARY OUTCOMES:
Pathological Response at the Time of Surgery | Weeks 10 to 28
  Specimen analysis according to TNM classification. Pathological complete response is defined as no invasive cancer cells in the surgical specimen.
R0 Resection rate at the Time of Surgery | Weeks 10 to 28
  The R0 resection rate after the neoadjuvant protocol. R0 is defined as a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed.
Tumor Regression Grade at the Time of Surgery | Weeks 10 to 28
  Estimate of tumor regression grade at the time of surgery according to Becker Criteria: Grade 1a, No residual tumor; Grade 1b, <10% residual tumor; Grade 2, 10-50% residual tumor; Grade 3, >50% residual tumor.
Lymph nodes response at the Time of Surgery | Weeks 10 to 28
  Participants were assessed for node-negative lymph nodes at the time of surgery according to TNM classification. Node-negative (pN0) participants had no regional lymph node metastasis.
Estimate of TN Change From Baseline to Surgery | Weeks 10 to 28
  Estimate of TN change due to neoadjuvant treatment is defined as the estimate of the evidence of downstaging between baseline and surgery

CONTACTS AND LOCATIONS:
Overall Officials: Javier Rodriguez Rodriguez, MD, PhD, Principal Investigator — Clinica Universidad de Navarra
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Background] Cunningham D, Allum WH, Stenning SP, Thompson JN, Van de Velde CJ, Nicolson M, Scarffe JH, Lofts FJ, Falk SJ, Iveson TJ, Smith DB, Langley RE, Verma M, Weeden S, Chua YJ, MAGIC Trial Participants. Perioperative chemotherapy versus surgery alone for resectable gastroesophageal cancer. N Engl J Med. 2006 Jul 6;355(1):11-20. doi: 10.1056/NEJMoa055531. PMID 16822992
- [Background] Xiong BH, Cheng Y, Ma L, Zhang CQ. An updated meta-analysis of randomized controlled trial assessing the effect of neoadjuvant chemotherapy in advanced gastric cancer. Cancer Invest. 2014 Jul;32(6):272-84. doi: 10.3109/07357907.2014.911877. Epub 2014 May 6. PMID 24800782
- [Background] Stahl M, Walz MK, Stuschke M, Lehmann N, Meyer HJ, Riera-Knorrenschild J, Langer P, Engenhart-Cabillic R, Bitzer M, Konigsrainer A, Budach W, Wilke H. Phase III comparison of preoperative chemotherapy compared with chemoradiotherapy in patients with locally advanced adenocarcinoma of the esophagogastric junction. J Clin Oncol. 2009 Feb 20;27(6):851-6. doi: 10.1200/JCO.2008.17.0506. Epub 2009 Jan 12. PMID 19139439
- [Background] Carton E, Caldwell MT, McDonald G, Rama D, Tanner WA, Reynolds JV. Specialized intestinal metaplasia in patients with gastro-oesophageal reflux disease. Br J Surg. 2000 Jan;87(1):116-21. doi: 10.1046/j.1365-2168.2000.01322.x. PMID 10606922
- [Background] Moehler M, Baltin CT, Ebert M, Fischbach W, Gockel I, Grenacher L, Holscher AH, Lordick F, Malfertheiner P, Messmann H, Meyer HJ, Palmqvist A, Rocken C, Schuhmacher C, Stahl M, Stuschke M, Vieth M, Wittekind C, Wagner D, Monig SP. International comparison of the German evidence-based S3-guidelines on the diagnosis and multimodal treatment of early and locally advanced gastric cancer, including adenocarcinoma of the lower esophagus. Gastric Cancer. 2015 Jul;18(3):550-63. doi: 10.1007/s10120-014-0403-x. Epub 2014 Sep 7. PMID 25192931
- [Background] Lee S, Oh SY, Kim SH, Lee JH, Kim MC, Kim KH, Kim HJ. Prognostic significance of neutrophil lymphocyte ratio and platelet lymphocyte ratio in advanced gastric cancer patients treated with FOLFOX chemotherapy. BMC Cancer. 2013 Jul 22;13:350. doi: 10.1186/1471-2407-13-350. PMID 23876227